CLINICAL TRIAL: NCT04933071
Title: Assessment of An Ob/Gyn Residency Podcast Curriculum on Resident Knowledge and Satisfaction
Brief Title: Ob/Gyn Residency Podcast Curriculum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Fei Cai, MD, Maternal Fetal Medicine Fellow, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 844674
Record Dates: First submitted 2021-06-13; First posted 2021-06-21 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Learning; Lack of (Specific); Medical Education
Keywords: Medical education; Graduate medical education; Obstetrics; Residency; Podcast

STUDY DESIGN:
Intervention Model Description: Residents in PGY-1 or PGY-2 group will be randomized to podcast learning (intervention) or usual teaching (no intervention)
Who Masked: Outcomes Assessor
Masking Description: Those that are grading residents (ie. attending physicians) will not be aware which arm the residents are randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Podcast Education (Experimental): Residents will be given access to podcasts during their rotation They will complete a survey after each obstetrics rotation
  Interventions: Behavioral: Podcast
- Usual Teaching (No Intervention): Residents will have usual teaching They will complete a survey after each obstetrics rotation

INTERVENTIONS:
Behavioral: Podcast — A list of podcasts that are specified for each rotation
  Arms: Podcast Education

SUMMARY:
This a randomized trial comparing the use of an organized podcast curriculum using the podcast, CREOGs Over Coffee, to usual teaching for first and second year Ob/Gyn residents on their obstetrics rotations. Residents at HUP and PAH will be included. Post intervention questionnaires will be administered at the end of each block to assess resident satisfaction with their block as well as confidence in their clinical care and skills. CREOG scores will be used to assess knowledge differences.

DETAILED DESCRIPTION:
All PGY-1 and PGY-2 Ob/Gyn residents at the Hospital of University of Pennsylvania (HUP) and Pennsylvania Hospital (PAH) will be eligible and recruited for this randomized trial over the period of January 2021 January 2023 (period chosen as CREOGs are given in January, and trial will start immediately after next CREOG exam). There are currently 7 PGY-1 residents and 8 PGY-2 residents at HUP and 7 PGY-1 residents and 8 PGY-2 residents at PAH. In two academic years, with the addition of 7 PGY-1 residents at HUP and 7 PGY-1 residents at PAH, this will total 43 residents.

Residents will be randomized individually to receive a podcast curriculum vs. usual teaching on the labor floor rotations. Rotations where there will be a podcast curriculum include labor and delivery, night float, and Maternal Fetal Medicine. The details of the curriculum for each rotation will be listed below. At all times, all residents will have access to the podcast content, but those randomized to usual teaching will not be given an organized podcast curriculum for each rotation. Currently, usual teaching includes didactic teaching for the above topics on Thursday mornings (7am-12 pm), clinical teaching while on the rotations, simulation training, and self-learning.

Residents will be protected against undue influence or coercion as those that are administering the surveys and recruiting residents (FC) will not be involved in their residency reviews.

ELIGIBILITY:
Inclusion Criteria:

* Residents that are PGY1-2 at the Hospital of the University of Pennsylvania and Pennsylvania Hospital in OB/Gyn

Exclusion Criteria:

* Those not meeting inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Resident Satisfaction | Week after rotation
  Satisfaction with rotation as seen on survey
Residence Confidence | Week after rotation
  Confidence in themselves as seen on survey

SECONDARY OUTCOMES:
CREOG Scores | January of each year within the study
  Scores based on percentiles of the CREOG (in-service exam) each year

CONTACTS AND LOCATIONS:
Overall Officials: Fei Cai, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No